CLINICAL TRIAL: NCT05199818
Title: Efficacy and Safety of Palonosetron HCl Buccal Film Versus IV Palonosetron for Prevention of Chemotherapy-induced Nausea and Vomiting in Cancer Patients Receiving Moderately Emetogenic Chemotherapy
Brief Title: Buccal Film vs IV Palonosetron for Prevention of CINV in Cancer Patients Receiving MEC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiamen LP Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LP-CT-PALO-202101
Record Dates: First submitted 2021-12-15; First posted 2022-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-08

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Palonosetron HCl Buccal Film (Experimental): Palonosetron HCl Buccal Film 0.5 mg 1 hr before administration of moderately emetogenic chemotherapy and normal saline injection 30 minutes before administration of moderately emetogenic chemotherapy
  Interventions: Drug: Palonosetron HCl Buccal Film 0.5 mg
- Palonosetron IV Injection (Active Comparator): Placebo buccal film 1 har before administration of moderately emetogenic chemotherapy and Palonosetron HCl Injection 0.25 mg 30 min before administration of moderately emetogenic chemotherapy
  Interventions: Drug: IV Palonosetron 0.25 mg

INTERVENTIONS:
Drug: Palonosetron HCl Buccal Film 0.5 mg — Palonosetron HCl Buccal Film and IV palonosetron placebo, both administered on Day 1
  Arms: Palonosetron HCl Buccal Film
Drug: IV Palonosetron 0.25 mg — IV Palonosetron and Palonosetron HCl Buccal Film placebo, both administered on Day 1
  Arms: Palonosetron IV Injection

SUMMARY:
The phase 3 study is to compare the efficacy and safety of palonosetron, a long-acting 5-HT3 receptor antagonist, by buccal film delivery compared to IV injection for the prevention of chemotherapy-induced nausea and vomiting. Subjects receive a single dose of palonosetron prior to moderately emetogenic chemotherapy.

DETAILED DESCRIPTION:
This is a phase 3 randomized, double-blind, parallel group study designed to evaluate the efficacy and safety of palonosetron HCL buccal film versus IV palonosetron for the prevention of chemotherapy-induced nausea and vomiting in cancer patients receiving moderately emetogenic chemotherapy (MEC).

Subjects are randomized into two treatment groups, one with the experimental study drug palonosetron in buccal film, the other one with the control treatment using Palonosetron hydrochloride IV injection. Palonosetron PK will be assessed in a subgroup of each treatment group (two sample points, 10% of subjects).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18-years of age;
2. Provide written informed consent;
3. Chemotherapy naïve subject with histologically or cytologically confirmed malignant disease; or chemotherapy non-naïve subject with histologically proven diagnosis of cancer;
4. Karnofsky index ≥ 50;
5. Be scheduled to receive MEC to be administered on Day 1;

Exclusion Criteria:

1. Unable to understand or cooperate with study procedure；
2. Received any investigational drug 30 days prior to study entry；
3. Used any drug with anti-emetic efficacy 24 hours prior to treatment and during the study；
4. Enrollment in a previous study with palonosetron；
5. Seizure disorder requiring anticonvulsant medication;
6. Experienced any vomiting, retching, or NCI Common Toxicity Criteria grade 2 or 3 nausea in the 24 hours preceding chemotherapy；
7. Ongoing vomiting from any organic etiology；
8. Experienced nausea (moderate to severe or vomiting following any previous chemotherapy)；
9. Scheduled to receive moderately or highly-emetogenic chemotherapy or radiotherapy during the study；
10. Known contraindication to 5-HT3 antagonist or dexamethasone；
11. Scheduled to receive bone marrow or stem cell transplant during study;
12. Symptomatic primary or metastatic CNS malignancy;
13. Lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Complete response | During the first 24 hours after chemotherapy
  No emetic episode and no rescue medication

SECONDARY OUTCOMES:
Complete response | 24-120 hours post chemotherapy
  No emetic episode and no rescue medication
Absence of nausea | up to 24 hours post chemotherapy, 24-120 hours post chemotherapy, and up to 120 hours post chemotherapy
  Absence of nausea based on daily patient questionnaire (yes or no) and no emetic episode or rescue medication
Complete response | up to 120 hours after chemotherapy
  The proportion of patients with complete response
Complete control | up to 24 hours post chemotherapy, 24-120 hours post chemotherapy, and up to 120 hours post chemotherapy
  The proportion of patients with complete control
Number of emetic episodes | up to 120 hours after chemotherapy
  Number of emetic episodes

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Pacific Cancer Medical Center, Anaheim, California
  - Watson Clinic, Lakeland, Florida
  - Lakes Research, Miami Lakes, Florida
  - Florida Cancer Affiliates, Ocala, Florida
  - Summit Cancer Care, Savannah, Georgia
  - Edward H. Kaplan MD & Associates, Skokie, Illinois
  - Orchard Healthcare research, Inc., Skokie, Illinois
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Tri-County Hematology & Oncology Associates, Massillon, Ohio
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania

IPD SHARING:
Plan to Share IPD: No